CLINICAL TRIAL: NCT05912764
Title: Evaluation of Early Home Return Care Pathway in Patients Who Have Undergone Endoscopic Enucleation of Prostate Adenoma by Laser
Brief Title: Evaluation of Early Home Return in Patients With Enucleation of Prostate Adenoma
Acronym: PRECODOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A00283-42
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Adenoma
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early home return arm (Experimental): Nurses will coordinate the patients' care prior to their intervention and when they leave the Clinics.
  Interventions: Other: Patient support
- Standard Of Care arm (No Intervention): Patients will not receive any support before and after intervention and hospital leave

INTERVENTIONS:
Other: Patient support — Patients will be supported by nurses before and after intervention and hospital leave
  Arms: Early home return arm

SUMMARY:
Prostate adenoma management includes, if necessary, surgical treatments: resection or vaporization by endoscopy or by open surgery in case of a very large prostate. Laser technology is a curative treatment for prostate adenoma. The minimum duration of hospitalization, in the context of enucleation prostatic endoscopy by laser, is estimated at 48 hours.

The Union Clinique has developed an improved rehabilitation care pathway reducing hospitalization duration to 24 hours (one night hospitalization). This care pathway involves patient as an actor in its care but also health professionals, in particular nurses.

This study is based on the hypothesis that the model developed by the Union Clinique can be translated to other healthcare establishments and that home return supervized by nurses allows reducing hospital stay length without increasing the risk of serious complications for patients

DETAILED DESCRIPTION:
Prostate adenoma management includes first drug treatments and, if necessary, surgical treatments: resection or vaporization by endoscopy or by open surgery in case of a very large prostate. Laser technology is a curative treatment for prostate adenoma. Its objective is to perform endoscopic excision (ablation) of the adenoma, in order to improve patients' quality of life and their urination. The laser energy is transmitted by a guided fiber under endoscopic control through the urethral canal in contact with the adenoma. Several wavelengths of the laser beam, depending on the nature of the generator crystals, are used for their specificity in cutting and tissue cauterization: Greenlight laser, Holmium laser, Thulium laser.

The minimum duration of hospitalization, in the context of an enucleation prostatic endoscopy by laser, is estimated at 48 hours. The Union Clinique has developed an improved rehabilitation care pathway reducing hospitalization duration to 24 hours (one night hospitalization). This care pathway involves patient as an actor in its care but also health professionals, in particular nurses, who will coordinate patients care prior to their intervention and when they leave the Clinics.

This study is based on the hypothesis that the model developed by the Union Clinique can be translated to other healthcare establishments and that home return supervized by health professionals, notably nurses, allows reducing hospital stay length without increasing the risk of serious complications for patients

ELIGIBILITY:
Inclusion Criteria:

* Patient planned for endoscopic enucleation of prostate adenoma with laser
* Patient with symptomatic benign prostatic hyperplasia and refractory to medical reatment and/or
* Patient with benign prostatic hyperplasia complicated by chronic retention of urine and/or
* Patient with benign prostatic hyperplasia complicated by prostatitis and/or
* Patient with symptomatic benign prostatic hyperplasia

Exclusion Criteria:

* Patient living beyond the scope of care by the nurses coordination
* Bedridden patient or WHO clinical condition >2
* Patient requiring curative anticoagulation which cannot be interrupted or relayed at home by heparin
* Patient with double anti-platelet aggregation who cannot be interrupted

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Re-hospitalizations and/or hospitalization extensions rate | 2 weeks
  the percentage of re-hospitalizations and/or hospitalization extensions

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROUVELLAT, MD, Principal Investigator — GCS RAMSAY SANTE
Locations (1):
- Clinique de l'Union, Saint-Jean, France

IPD SHARING:
Plan to Share IPD: No